CLINICAL TRIAL: NCT02789813
Title: Randomized Placebo-controlled Phase II Study on the Influence of Valproic Acid in Combination With Reactivation of Fear Memory on the Outcome of Extinction-based Therapy in Patients With Fear of Spiders.
Brief Title: Influence of Valproic Acid on Extinction-based Therapy in Patients With Fear of Spiders.
Acronym: VALPRO
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Prof. Dominique de Quervain, MD (Other)
Responsible Party: Sponsor-Investigator, Prof. Dominique de Quervain, MD, MD, University of Basel
Organization: University of Basel (Other)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 2016DR2001
Record Dates: First submitted 2016-04-20; First posted 2016-06-03 (Estimated); Last update posted 2018-10-02 (Actual); Status verified 2018-10

CONDITIONS: Phobia, Specific
MeSH Terms: conditions — Phobia, Specific | interventions — Valproic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (4):
- Valproic Acid and fear reactivation (Experimental): This group will receive once a combination of 500mg Valproic Acid (oral solution) and fear reactivation before exposure therapy.
  Interventions: Drug: Valproic Acid; Behavioral: Fear reactivation
- Valproic Acid and no fear reactivation (Active Comparator): This group will receive once 500mg Valproic Acid (oral solution) before exposure therapy.
  Interventions: Drug: Valproic Acid; Behavioral: No fear reactivation
- Placebo and fear reactivation (Placebo Comparator): This group will receive once a combination of Placebo (oral solution) and fear reactivation before exposure therapy.
  Interventions: Drug: Placebo; Behavioral: Fear reactivation
- Placebo and no fear reactivation (Placebo Comparator): This group will receive once Placebo (oral solution) before exposure therapy.
  Interventions: Drug: Placebo; Behavioral: No fear reactivation

INTERVENTIONS:
Drug: Valproic Acid — Once oral administration of 500mg before exposure therapy.
  Other Names: Orfiril®
  Arms: Valproic Acid and fear reactivation; Valproic Acid and no fear reactivation
Drug: Placebo — Once oral administration of 500mg before exposure therapy.
  Arms: Placebo and fear reactivation; Placebo and no fear reactivation
Behavioral: Fear reactivation — Fear reactivation before exposure therapy.
  Arms: Placebo and fear reactivation; Valproic Acid and fear reactivation
Behavioral: No fear reactivation — No fear reactivation before exposure therapy.
  Arms: Placebo and no fear reactivation; Valproic Acid and no fear reactivation

SUMMARY:
The purpose of this study is to evaluate whether valproic acid in combination with fear memory reactivation is useful to enhance treatment stability of exposure therapy for specific phobia.

DETAILED DESCRIPTION:
* There will be one screening visit (visit 1), one intervention visit (visit 2) and one follow-up visit (90 days after visit 2) (visit 3).
* On visit 2 all participants will undergo 30 min exposure therapy in virtual reality with pre-defined spider situations.
* Duration for an individual participant will be at most 15 weeks depending on the time passing between screening (visit 1) and intervention visit (visit 2).
* Change in phobic fear to baseline (visit 1) will be assessed on 90 day follow-up (visit 3).
* Documentation of all study relevant source data of every study participant will be done by completing the study specific electronic case report forms (eCRF, SoSci Survey) and study specific case report forms on paper (Adverse Events, Serious Adverse Events and concomitant medication). Data in the eCRF can be validated for completeness and discrepancies automatically. An audit trail system maintains a record of initial entries and changes (reasons for changes, time and date of changes, user identification of entry and changes).
* Quality insurance will be done by an external site monitoring (including study progress, accuracy and completeness of eCRF, fulfillment of protocol requirements, applicable local authority regulations and investigator's obligations).
* Monitoring includes 100% of safety parameters, primary endpoints, informed consent documents and the Trial Master File on the Initiation Visit and on Close Out.
* Standard Operating Procedures to address study activities such as patient recruitment, informed consent, study interventions, data collection, data management, data analysis, and reporting for adverse events exist.

ELIGIBILITY:
Inclusion Criteria:

* DSM-IV diagnosis of specific phobia (animal type: spider)
* BAT score (at screening) between 1 and 7 points
* Physically healthy
* Normotensive (90/60-140/90 mmHg)
* Male or female
* Aged between 18 and 40 years
* Native or fluent German-speaking
* Females have to be on effective birth control

Exclusion Criteria:

* Other axis I disorder except a further comorbid phobic disorder
* Concurrent psychotherapy or pharmacotherapy
* Previous exposure-based therapy for specific phobia
* Parallel participation in another study
* Body weight less than 50kg
* Long-term medication intake
* Substance abuse
* 5 or more cigarettes a day and/or inability of being abstinent for at least 5 hours
* Pregnancy or breast-feeding
* Kinetosis
* History of coagulation disease
* History of gastrointestinal disease
* Laboratory exclusion criteria: clinically relevant deviation of laboratory values (blood count, blood chemistry, coagulation status, liver and pancreas enzymes, electrolytes) from normal range

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 100 (Actual)
Dates: Start 2016-07; Primary Completion 2018-06-30 (Actual); Study Completion 2018-06-30 (Actual)

PRIMARY OUTCOMES:
Change in performance in Behavioral Approach Test (BAT) in real-life (in vivo) | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention

SECONDARY OUTCOMES:
Change in performance in BAT in virtual reality (in virtuo) | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention
Change in subjective reactions in BAT in virtual reality (in virtuo) | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention
Change in psychophysiological reactions in BAT in virtual reality (in virtuo) | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention
Change in subjective reactions to fear-related picture cue presentation quantified by visual analog scales (VAS) for valence, arousal and fear | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention
Change in psychophysiological reactions to fear-related picture cue presentation quantified by electrodermal activity (EDA), heart rate (HR), startle response | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention
Performance in working and recognition memory of pictures task | Follow up (visit 3: 90 days after visit 2: intervention)
Valence, arousal, and mood ratings of pictures of working and recognition memory of pictures task | Follow up (visit 3: 90 days after visit 2: intervention)
Change in strength of phobic fear quantified by self-report questionnaires | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)
Change in mood and state-anxiety quantified by self-report questionnaires | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)
Change in performance during exposure in virtuo quantified by eye tracking | Intervention (visit 2: 7-21 days after visit 1: baseline)
Change in subjective reactions during exposure in virtuo quantified by subjective units of discomfort (SUD) ratings | Intervention (visit 2: 7-21 days after visit 1: baseline)
Change in psychophysiological reactions during exposure in virtuo quantified by EDA and HR | Intervention (visit 2: 7-21 days after visit 1)
Change in clinical relevance of phobic symptoms measured by Diagnostic Interview for Psychiatric Disorders (DIPS), section for specific phobia | Baseline (visit 1: 7-21 days before visit 2: intervention) and follow up (visit 3: 90 days after visit 2: intervention)

OTHER OUTCOMES:
Adverse Events | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)
Blood pressure | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)
Heart rate | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)
VAS of headache, stomach pain, nausea, fatigue, dizziness, drowsiness muscle fatigue, and motivation. | Baseline (7-21 days before visit 2: intervention), intervention (visit 2: 7-21 days after visit 1: baseline) and follow up (visit 3: 90 days after visit 2: intervention)

CONTACTS AND LOCATIONS:
Overall Officials: Dominique JF de Quervain, MD, Principal Investigator — University of Basel
Locations (1):
- Psychiatric University Clinics, University Basel, Basel, Switzerland

IPD SHARING:
Plan to Share IPD: No